CLINICAL TRIAL: NCT03567577
Title: Safety and Preliminary Efficacy of Sequential Multiple Ascending Doses of Solnatide to Treat Pulmonary Permeability Oedema in Patients With Moderate-to-severe ARDS - a Randomised, Placebo-controlled, Double-blind Trial
Brief Title: Safety and Preliminary Efficacy of Sequential Multiple Ascending Doses of Solnatide to Treat Pulmonary Permeability Oedema in Patients With Moderate-to-severe ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apeptico Forschung und Entwicklung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP301-II-002
Record Dates: First submitted 2018-04-23; First posted 2018-06-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: ARDS
Keywords: Peptide
MeSH Terms: interventions — AP301 peptide; Powders; Solutions; Inhalation; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Solnatide 5mg (Experimental): Solnatide 25 mg powder for reconstitution for solution for inhalation. 5mg administered
  Interventions: Drug: Solnatide 25 mg powder for reconstitution for solution for inhalation
- Solnatide 60mg (Experimental): Solnatide 25 mg powder for reconstitution for solution for inhalation. 60mg administered
  Interventions: Drug: Solnatide 25 mg powder for reconstitution for solution for inhalation
- Solnatide 125mg (Experimental): Solnatide 25 mg powder for reconstitution for solution for inhalation. 125mg administered
  Interventions: Drug: Solnatide 25 mg powder for reconstitution for solution for inhalation
- Placebo (Placebo Comparator): 0,9% saline solution
  Interventions: Drug: 0.9% Saline Solution

INTERVENTIONS:
Drug: Solnatide 25 mg powder for reconstitution for solution for inhalation — Inhalation of an aerosol every 12 hours (± 30 min), for a total of 7 days.
  Other Names: AP301
  Arms: Solnatide 125mg; Solnatide 5mg; Solnatide 60mg
Drug: 0.9% Saline Solution — Inhalation of an aerosol every 12 hours (± 30 min), for a total of 7 days.
  Arms: Placebo

SUMMARY:
This phase IIb, randomized, placebo-controlled, double-blind, dose escalation study will assess the local and systemic safety of 7 days orally inhaled sequential multiple ascending doses of solnatide in patients with pulmonary permeability oedema and moderate-to-severe ARDS and review potential efficacy endpoints for a future phase III pivotal trial.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Male or female ≥18 years of age.
3. Patient has been admitted to an ICU, is mechanically ventilated (according to the ventilation and weaning protocol in Appendix I) and stable in this condition for at least 8 hours.
4. Moderate-to-severe ARDS diagnosis as defined by the Berlin Definition:

   * Onset of ARDS within 1 week of a known clinical insult or new or worsening respiratory symptoms.
   * Bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules.
   * Respiratory failure not fully explained by cardiac failure or fluid overload (origin of oedema).
   * PaO2/FiO2 ≤ 200 mm Hg with Positive End-Expiratory Pressure (PEEP) ≥5 cm H2O.
5. ARDS diagnosis not older than 48 hours.
6. Extravascular lung water index (EVLWI) ≥ 10 ml/PBW as assessed with a validated bedside measurement (single indicator transpulmonary thermodilution measurement with the PiCCO® system).
7. Patient who meets criteria for extensive hemodynamic monitoring as per international intensive care medicine standards.
8. For patients that are temporarily unable to consent (e.g. comatose patients) a subsequent informed consent has to be provided.
9. Male and Female (WOCBP) patients using adequate contraception.

Exclusion Criteria:

1. History of clinically relevant allergies or idiosyncrasies to solnatide.
2. Known use of any other investigational or non-registered drug within 30 days prior to study enrolment.
3. Severe state of septic shock with a Mean Arterial Pressure (MAP) ≤ 65 mm Hg and a serum lactate level > 4 mmol/L (36 mg/dL) despite adequate volume resuscitation.
4. An underlying clinical condition that, in the opinion of the Investigator, would make it very unlikely for the patient to be successfully weaned from ventilation due to severe underlying diseases (e.g. severe malnutrition, severe neurological diseases, pulmonary fibrosis or COPD).
5. Extra-corporeal membrane oxygenation, high-frequency oscillatory ventilation or any form of extra-corporeal lung support. In no way are patients to be denied or delayed these procedures to avoid exclusion from the study.
6. Neutrophil count < 0.3 x 109/L.
7. Cancer treatment (chemotherapy or biological) or therapy with other immunosuppressive agents for organ transplantation within 2 weeks.
8. Cachexia (BMI < 18.5 kg/m2).
9. Cardiogenic pulmonary oedema diagnosed by echocardiography or pulmonary artery catheter.
10. Severe skin burns involving more than 15% of body surface.
11. Subjects who are extremely unlikely to survive more than 48 hours due to the acute conditions of the patient in the opinion of the Investigator.
12. Subjects transferred from a hospital not participating in this study who are already planned to be re-transferred during the observation period.
13. Subjects who are not expected to survive the next month because of an underlying uncorrectable medical condition or a do not resuscitate order.
14. Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Safety endpoint: Any cause death | Randomisation - day 28
  Primary Safety Endpoint: Composite endpoint including any cause death at day 28
Safety endpoint: Drug-related adverse events | Randomisation - day 14
  Primary Safety Endpoint: Composite endpoint including drug-related adverse events through day 14
Safety endpoint: All adverse events | Randomisation - day 28
  Primary Safety Endpoint: Composite endpoint including all adverse events through day 28

SECONDARY OUTCOMES:
EVLWI | baseline - day 7
  Change in extravascular lung water index (EVLWI) as assessed with a validated bedside measurement (measurement with the PiCCO® system)
PVPI | baseline - day 7
  Change in pulmonary vascular permeability index (PVPI) as assessed with a validated bedside measurement (measurement with the PiCCO® system)
Change of ventilatory settings | baseline - day 14
  Composite endpoint including ventilation mode, ventilation pressures (ventilatory plateau pressure, positive end expiratory pressure, peak inspiratory pressure, mean airway pressure, peak airway pressure, driving pressure), tidal volume
Murray lung injury score | baseline - day 7
  Murray lung injury score is composed of four components: 1) chest radiograph; 2) hypoxaemia score; 3) PEEP and 4) static compliance of respiratory system. The values of the total score may range from 0 to 4. Lower values indicate a better outcome.
Oxygenation ratio (PaO2 / FiO2 ratio) | baseline - day 7
Time to extubation | baseline - day 28
Ventilator-free days (VFD) | baseline - day 28
Days of hospitalization and in ICU | baseline - day 28

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (3):
  - Univ.-klinik f. Herz-, Thorax-, Gefäßchirurgische Anästhesiologie und lntensivmedizin, Medizinische Universität Graz, Graz, Styria
  - Department of Anesthesia, General Intensive Care and Pain Control,Medical University of Vienna, Vienna, Vienna
  - Univ. Klinik für Innere Medizin / Gem. Einrichtung für Intensiv- und Notfallmedizin/GE Medizinische Universität Innsbruck, Innsbruck
- Germany (12):
  - Klinik für Anaesthesiologie, Klinikum der Universität München, Campus Großhadern, München, Bavaria
  - Klinik für Operative Intensivmedizin und Intermediate Care, Aachen, North Rhine-Westphalia
  - Klinik und Poliklinik für Anästhesiologie und Intensivtherapie / Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Bonn, Operative Intensivmedizin, Klinik und Poliklinik für Anästhesiologie und Operative Intensivmedizin, Bonn
  - Georg-August-Universität Göttingen, Göttingen
  - Klinik für Anästhesiologie und operative Intensivmedizin, Universitätsklinikum Schleswig-Holstein, Campus Kiel,, Kiel
  - Klinik für Anästhesiologie / Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinik für Anästhesiologie und operative Intensivmedizin; Universitätsmedizin Mannheim, Mannheim
  - Klinik für Anästhesiologie und Intensivmedizin; Klinikum rechts der Isar der TU München, München
  - Klinik und Poliklinik für Innere Medizin II; Klinikum rechts der Isar der TU München, München
  - Klinik für Anästhesiologie, operative Intensivmedizin und Schmerztherapie; Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Klinik und Poliklinik für Anästhesiologie, Würzburg

IPD SHARING:
Plan to Share IPD: No